CLINICAL TRIAL: NCT01020305
Title: Temsirolimus, an mTOR Inhibitor, to Reverse Androgen Insensitivity in Patients With Castration-resistant Prostate Cancer
Brief Title: Temsirolimus to Reverse Androgen Insensitivity for Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision by funding sponsor due to poor accrual
Sponsor: Sandy Srinivas (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); National Comprehensive Cancer Network (Network); American Society of Clinical Oncology (Other)
Responsible Party: Sponsor-Investigator, Sandy Srinivas, Assoc Prof-Med Ctr Line, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17242; NCT01020305 (Other: NIH); SU-09292009-4080 (Other: Stanford University); PROS0028 (Other: OnCore)
Record Dates: First submitted 2009-10-30; First posted 2009-11-25 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Castrate-resistant Prostate Cancer (CRPC); Androgen-insensitive Prostate Cancer; Hormone-refractory Prostate Cancer; Metastatic Disease
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — temsirolimus; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus + Bicalutamide (Experimental): Temsirolimus 25 mg administered intravenously (IV) once weekly for 12 weeks
  Casodex (bicalutamide) administered 50 mg/day orally (PO)
  Interventions: Drug: Temsirolimus; Drug: Casodex (bicalutamide)

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus is an inhibitor of the mammalian target of rapamycin (MTOR, aka HGNC:3942)
  IUPAC name: (1R,2R,4S)-4-{(2R)-2-[(3S,6R,7E,9R,10R,12R,14S,15E,17E,19E,21S,23S,26R,27R,34aS)-9,27-dihydroxy-10,21-dimethoxy-6,8,12,14,20,26-hexamethyl-1,5,11,28,29-pentaoxo-1,4,5,6,9,10,11,12,13,14,21,22,23,24,25,26,27,28,29,31,32,33,34,34a-tetracosahydro-3H-23,27-epoxypyrido[2,1-c][1,4]oxazacyclohentriacontin-3-yl]propyl}-2-methoxycyclohexyl 3-hydroxy-2-(hydroxymethyl)-2-methylpropanoate
  Other Names: Torisel; CCI-779
Drug: Casodex (bicalutamide) — Casodex (bicalutamide) 50 mg/day PO
  Other Names: Casodex; bicalutamide; Cosudex; Calutide; Kalumid

SUMMARY:
This study evaluates if temsirolimus causes a reduction in the serum levels of prostate-specific antigen (PSA) in male subjects with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
Castration-resistant prostate cancer (CRPC) is also known as "androgen-insensitive" or "hormone-refractory" prostate cancer. While numerous therapies impact biochemical response in the setting of CRPC, there remains unmet medical need. New therapies that extend survival of patients beyond that provided by chemotherapy are needed.

The mechanisms of tumor progression to castration-resistance are unclear, but preclinical studies suggest that functional loss of the tumor suppressor gene PTEN and subsequent up-regulation of Akt, which is upstream of mTOR, may be involved in prostate cancer progression and metastasis. Based on these observations, it is hypothesized that mTOR inhibitor temsirolimus may prolong hormone sensitivity and delay disease progression in castration-resistant prostate cancer patients before antiandrogen withdrawal.

This study will assess efficacy on the basis of serum levels of PSA, an established surrogate endpoint for efficacy in prostate cancer.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically-confirmed adenocarcinoma of the prostate, characterized as symptomatic castration-resistant prostate cancer (CRPC)
* Serum PSA ≥ 2 ng/mL
* Rising PSA on 3 consecutive occasions at least 1 week apart (not limited to the 30-day screening period)
* Failure of bilateral orchiectomy and/or therapy with an LHRH agonist and bicalutamide
* Castrate level of testosterone (< 50 ng/dL)
* Currently being treated with bicalutamide
* No prior antiandrogen therapy except bicalutamide
* Age ≥ 18 years
* Life expectancy > 6 months
* Performance status

  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
  * OR
  * Karnofsky performance status ≥ 80%
* Ability to understand and the willingness to sign a written informed consent

EXCLUSION CRITERIA

* Radiotherapy for prostate cancer within 28 days prior to Day 1, except single-fraction radiotherapy for pain control
* Prior treatment with mTOR inhibitors
* Prior treatment with chemotherapy for prostate cancer
* Symptomatic bone metastases (ie, asymptomatic bone metastases are eligible)
* Visceral metastases
* Absolute neutrophil count (ANC) < 1500/uL
* Platelet count ≤ 100 x 10e9/L
* Total bilirubin ≥ 1.5 x Upper Limit of Normal (ULN)
* Alkaline phosphatase > 2.5 x ULN
* AST > 2.5 x ULN
* ALT > 2. 5x ULN
* Serum creatinine > 2.0 mg/dL
* Hemoglobin < 9 g/dL
* Men with reproductive potential who do not agree to use an accepted and effective method of contraception during the study treatment period and for at least 3 months after completion of the study treatment
* History of other malignancies within 5 years except for tumors with a negligible risk for metastasis or death, such as adequately-controlled basal cell carcinoma, squamous-cell carcinoma of the skin, or early-stage bladder cancer
* Participation in another experimental drug study either planned or within 4 weeks of the first study treatment
* Persistent Grade ≥ 1 AEs due to prior drug therapy, including investigational drugs, administered more than 14 days before study enrollment
* Previously treated or other known brain metastases
* Ongoing or active infection
* Symptomatic congestive heart failure, New York Heart Association Grade II or greater
* Unstable angina pectoris
* Cardiac arrhythmia
* Significant vascular disease (eg, aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Psychiatric illness/social situations that would limit compliance with study requirements
* Other uncontrolled intercurrent illness
* Known to be positive for the human immunodeficiency virus (HIV) infection and receiving antiretroviral therapies (HIV positive not requiring antiretroviral therapy iseligible if all other entry criteria are meet)
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya "Sandy" Srinivas, MD, Principal Investigator — Stanford University; Lauren Christine Harshman, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Temsirolimus + Bicalutamide: Temsirolimus 25 mg administered intravenously (IV) once weekly for 12 weeks
  Casodex (bicalutamide) administered 50 mg/day orally (PO)
  Temsirolimus: Temsirolimus is an inhibitor of the mammalian target of rapamycin (MTOR, aka HGNC:3942)
  IUPAC name: (1R,2R,4S)-4-{(2R)-2-[(3S,6R,7E,9R,10R,12R,14S,15E,17E,19E,21S,23S,26R,27R,34aS)-9,27-dihydroxy-10,21-dimethoxy-6,8,12,14,20,26-hexamethyl-1,5,11,28,29-pentaoxo-1,4,5,6,9,10,11,12,13,14,21,22,23,24,25,26,27,28,29,31,32,33,34,34a-tetracosahydro-3H-23,27-epoxypyrido[2,1-c][1,4]oxazacyclohentriacontin-3-yl]propyl}-2-methoxycyclohexyl 3-hydroxy-2-(hydroxymethyl)-2-methylpropanoate
  Casodex (bicalutamide): Casodex (bicalutamide) 50 mg/day PO
Period: Overall Study
Arm/Group | Temsirolimus + Bicalutamide
Started | 5
Completed | 3
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Temsirolimus + Bicalutamide
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 73 [64 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Serum PSA
Description: Proportion of subjects with > 50% drop in serum PSA as compared to baseline, assessed at 16 weeks
Time Frame: 12 weeks treatment, with primary outcome assessed at 16 weeks
Measure: Number; unit: participants
Arm/Group | Temsirolimus + Bicalutamide
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Arm/Group | Temsirolimus + Bicalutamide
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus + Bicalutamide (N=5)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temsirolimus + Bicalutamide (N=5)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Other-Tachycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Edema, trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Other-fall (General disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 3 (3)
Increase ALT (Investigations) | 2 (2)
Increase AST (Investigations) | 2 (2)
Increase creatinine (Investigations) | 2 (2)
Increase in HDL (Investigations) | 2 (2)
Increase LDL (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Other-Bilateral Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other-Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No